CLINICAL TRIAL: NCT00134511
Title: Phase 3 Multi-Center, Open Label, Forced Titration Study To Evaluate The Efficacy, Safety, And Tolerability Of Torcetrapib/Atorvastatin Combination Administered Orally, Once Daily (Qd) In Patients With Homozygous Familial Hypercholesterolaemia
Brief Title: Study To Evaluate The Effect Of Torcetrapib/Atorvastatin In Patients With Genetic High Cholesterol Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A5091027
Record Dates: First submitted 2005-08-22; First posted 2005-08-24 (Estimated); Last update posted 2007-11-07 (Estimated); Status verified 2006-12

CONDITIONS: Hypercholesterolemia, Familial
MeSH Terms: conditions — Hyperlipoproteinemia Type II | interventions — torcetrapib; Atorvastatin

INTERVENTIONS:
Drug: Torcetrapib/atorvastatin

SUMMARY:
The Torcetrapib project was terminated on December 2, 2006 due to safety findings.

To evaluate the efficacy and safety of the lipid drug Torcetrapib/atorvastatin in patients with genetically known disorder of extremely high cholesterol

DETAILED DESCRIPTION:
For additional information please call: 1-800-718-1021

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Homozygous Familial Hypercholesterolemia

Exclusion Criteria:

* Women who are pregnant or lactating, or planning to become pregnant.
* Subjects with a clinically indicated need for statin (HMG-CoA reductase inhibitor) therapy other than atorvastatin or other concomitant therapy with known lipid altering effects on LDL-C and HDL-C including fibrates and nicotinic acid
* Subjects taking any drugs known to be associated with an increased risk of myositis in combination with HMG-CoA reductase inhibitors
* Subjects with any other medical condition or laboratory abnormality which could affect subject safety, preclude evaluationof response, or render unlikely that the subject would complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2005-03; Study Completion 2005-11

PRIMARY OUTCOMES:
Change in LDL-C and HDL-C

SECONDARY OUTCOMES:
Other lipid variables

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- Pfizer Investigational Site, Boston, Massachusetts, United States
- Canada (2):
  - Pfizer Investigational Site, Chicoutimi, Quebec
  - Pfizer Investigational Site, Ste-Foy, Quebec
- South Africa (3):
  - Pfizer Investigational Site, Parktown, Johannesburg
  - Pfizer Investigational Site, Bloemfontein
  - Pfizer Investigational Site, Cape Town